CLINICAL TRIAL: NCT00808535
Title: A Pilot Study of Cardiac Magnetic Resonance Imaging For Detection of Myocardial Perfusion Abnormalities in Endothelial Dysfunction
Brief Title: Cardiac Magnetic Resonance Imaging for Detecting Endothelial Dysfunction
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of California, Los Angeles (Other)
Collaborators: Bracco Diagnostics, Inc (Industry)
Responsible Party: Stefan Ruehm, MD, UCLA
Other Study IDs: CMRI_Perfusion Study
Record Dates: First submitted 2008-12-15; First posted 2008-12-16 (Estimated); Last update posted 2009-02-09 (Estimated); Status verified 2009-02

CONDITIONS: Endothelial Dysfunction; Myocardial Perfusion Abnormalities; Cardiac MRI Perfusion With Vasomotor Stress; Diabetes
Keywords: Endothelial dysfunction; Cardiac Perfusion MRI; Vasomotor Stress; Cold Pressor Test; Adenosine Stress
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- diabetics
  Interventions: Procedure: Cardiac Perfusion MRI w Vasomotor Stress
- healthy controls
  Interventions: Procedure: Cardiac Perfusion MRI w Vasomotor Stress

INTERVENTIONS:
Procedure: Cardiac Perfusion MRI w Vasomotor Stress — All participants will undergo Cardiac Perfusion MRI with Vasomotor Stress. Vasomotor Stress will include both Cold Pressor Test and Adenosine Stress Test.

SUMMARY:
The goal of this research study is to demonstrate that Cardiac Perfusion MRI with Vasomotor Stress may serve as a non-invasive and less risky imaging technique for detecting non-obstructive perfusion deficits and/or abnormalities in myocardial blood flow (MBF) in patients with endothelial dysfunction.

This is a controlled study, which will enroll approximately 60 subjects (30 diabetics and 30 non-diabetics to serve as healthy controls), and will include male and non-pregnant females, between the ages 18-50 years.

All eligible participants will sign an informed consent and will complete a Lifestyle Questionnaire. They will undergo blood work which includes:

* 2-hour Oral Glucose Tolerance Test and Fasting Labs for Glucose, Insulin, C-Peptide, HbA1c, Creatinine, and Lipid Panel.
* Urine Albumin to Creatinine ratio for microalbuminuria.
* Serum inflammatory markers: E-selectin, homocysteine, ADMA, VCAM, IL-6, TNFalpha, hs-CRP and PAI-1.

After blood work, all participants will undergo cardiac MR perfusion imaging procedure with Cold Pressor Test and Adenosine Stress Test.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 50 years
* Should be able to sign an informed consent and HIPAA Agreement
* 30 healthy, non-diabetic individuals
* 30 diabetic individuals without documented coronary artery disease
* Diagnosed diabetics less than 5 years
* HbA1c less than 8.0

Exclusion Criteria:

* Children under 18 years and adults above 50 years
* Type 1 DM
* Lactating and Pregnant females
* BMI less than 35
* Contraindication to MRI such as pacemaker, defibrillator implants, etc.
* Allergy to MR (paramagnetic) contrast
* History of Angina, MI, or documented Coronary Artery Disease
* Previous history of CHF, CABG, Angioplasty and Stenting
* History of Valvular Heart Disease and Congenital Heart Disease
* History of Peripheral Vascular Disease
* History of Cardiac Arrythmias and anti-coagulation therapy
* History of Cerebro-vascular accidents or TIA
* History of active diabetic retinopathy and nephropathy
* Uncontrolled hypertension (systolic > 170 and diastolic >100 mm Hg
* End Stage Renal Disease and patients on dialysis
* HbA1c of 8.0
* Creatinine greater than 1.7 mg/dl
* History of active gastrointestinal bleeding
* History of IV drug use
* Chronic or current steroid treatment
* Growth hormone treatment

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Diagnosed diabetics (less than 5 years) without documented coronary artery disease recruited from UCLA Ambulatory clinics.
  Healthy controls from general population.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2009-02; Primary Completion 2010-02 (Estimated); Study Completion 2010-03 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Ruehm, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Radiological Sciences, Los Angeles, California, United States